CLINICAL TRIAL: NCT00151463
Title: An Open-Label, Non-Comparative Study To Evaluate Treatment Responsiveness To The Quality Of Erection Questionnaire (QEQ) In Men With Erectile Dysfunction Treated With Viagra (Sildenafil Citrate)
Brief Title: QEQ Treatment Responsiveness Evaluation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481195
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil citrate

SUMMARY:
The Quality of Erection Questionnaire (QEQ) is a new questionnaire that was developed to assess erectile attributes in men with erectile dysfunction. The study objective is to validate the Quality of Erection Questionnaire (QEQ) through the evaluation of subject responses to the QEQ regarding the quality and hardness of erections at baseline compared to subject responses post 6 and 10 weeks dosing with Viagra (sildenafil citrate).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented clinical diagnosis of erectile dysfunction based on a screening SHI-M score of <21 and the subject fulfilling the NIH definition of erectile dysfunction
* Subjects must be either PDE-5 inhibitor naive; i.e. have never used sildenafil, tadalafil or vardenafil, or have been previously treated with no more than six doses of a PDE-5 inhibitor (sildenafil, tadalafil, vardenafil) and must have taken their last dose no less than 4 weeks prior to the screening visit

Exclusion Criteria:

* Subjects who are currently prescribed, taking and/or likely to be treated with nitrates or nitric oxide donors in any form on either a regular or intermittent basis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01

PRIMARY OUTCOMES:
Treatment response to the Quality of Erection Questionnaire (QEQ) after treatment with Viagra in men with erectile dysfunction

SECONDARY OUTCOMES:
Change from baseline to week 6 of the QEQ total score
Change from baseline to week 6 in the 5 IIEF domain scores
Change from baseline in scores of QEQ individual question

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Australia (9):
  - Pfizer Investigational Site, Bondi Junction, New South Wales
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Spring Hill, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Malvern, Victoria
  - Pfizer Investigational Site, Mentone, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481195&StudyName=QEQ+Treatment+Responsiveness+Evaluation+Study